CLINICAL TRIAL: NCT02696850
Title: The Impact Of The Addition Of Budesonide To Low-Pressure, High-Volume Saline Sinus Irrigation For Chronic Rhinosinusitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201512063
Record Dates: First submitted 2016-02-26; First posted 2016-03-02 (Estimated); Results first posted 2019-09-03 (Actual); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Rhinosinusitis; Chronic Eosinophilic Rhinosinusitis; Allergic Rhinosinusitis
Keywords: sinusitis; rhinosinusitis; rhinitis; nasal lavage
MeSH Terms: conditions — Rhinosinusitis; Rhinitis, Allergic, Perennial; Sinusitis; Rhinitis | interventions — Budesonide; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Budesonide (Experimental): The study intervention will be budesonide powder (0.5 mg/capsule). Subjects will be required to dissolve the contents of two capsules into the 8-ounce (240 ml) NeilMed Sinus Rinse Regular Bottle along with the saline rinse. All subjects will be instructed to irrigate both right and left nasal cavity with one-half of the contents of the nasal rinse once daily.
  Each study bottle will contain 60 capsules of Budesonide and will be assigned with a number from 1-80.
  Interventions: Drug: Budesonide
- Saline Alone (Placebo Comparator): Each study bottle will contain 60 capsules of placebo, which is lactose monohydrate and will be supplied in clear plastic capsules identical to the budesonide capsules. Subjects will be required to dissolve the contents of two capsules into the 8-ounce (240 ml) NeilMed Sinus Rinse Regular Bottle along with the saline rinse. All subjects will be instructed to irrigate both right and left nasal cavity with one-half of the contents of the nasal rinse once daily.
  Interventions: Drug: Saline alone

INTERVENTIONS:
Drug: Budesonide — Participants will undergo 4-week treatment course that includes budesonide powder added to saline rinse.
  Arms: Budesonide
Drug: Saline alone — Participants will undergo 4-week treatment course that includes lactose (placebo) powder added to saline rinse.
  Arms: Saline Alone

SUMMARY:
The goal of this research project is to explore the impact of the addition of budesonide to high-volume, low-pressure nasal sinus saline irrigation (aka "Neti-Pot"-type systems) for patients with chronic rhinosinusitis with or without nasal polyps.

DETAILED DESCRIPTION:
Study Design

Double-blind placebo-controlled randomized clinical trial

Subjects Up to 80 adult patients with complaints of purulent (not clear) nasal drainage accompanied by nasal obstruction, facial pain-pressure-fullness, or both and reduction or loss of smell for 12 weeks or greater.

Inclusion Criteria:

Twelve (12) weeks or longer of two or more of the following signs and symptom consistent with chronic rhinosinusitis (CRS):

mucopurulent drainage (anterior, posterior, or both), nasal obstruction (congestion),facial pain-pressure-fullness, and decreased sense of smell

AND inflammation documented by one or more of the following findings:

* purulent (not clear) mucus or edema in the middle meatus or ethmoid region,
* polyps in nasal cavity or the middle meatus, and/or
* radiographic imaging showing inflammation of the paranasal sinuses

Exclusion criteria:

* Unable to speak English
* History of comorbid ciliary dyskinesia, cystic fibrosis or any other mucociliary condition
* Dependence on prolonged corticosteroid therapy for comorbid condition, such as asthma and chronic obstructive pulmonary disease.
* History of oral or systematic antibiotic use in the past 2 weeks
* History of nasal or sinus surgery within past 6 weeks
* History of cerebrospinal fluid leak
* History of allergy to budesonide or other topical steroids
* Pregnant or breast feeding
* Current infection or history of one of the following infections: Tuberculosis (TB) lung infection, or Herpes infection of the eye.
* Baseline SNOT-22 total scores below 9 were excluded due to the inability to achieve a minimally clinically improved difference

Variables of Interest Demographic - age, gender, and race. Index condition - Duration of CRS symptoms, response to previous treatments Co-morbid conditions - Presence and severity of general comorbid conditions will be assessed with ACE-27. Presence of rhinosinusitis-specific comorbidities will include: inhalant allergies, asthma, and aspirin sensitivity Previous sinus and/or nasal surgery - Previous sinus and/or nasal surgery, including functional endoscopic sinus surgery, turbinate reduction, and septoplasty will be captured and duration since surgery to time of enrollment.

Randomization The study statistician, Dr. Dorina Kallogjeri, will use a randomized block design for study drug assignment. To ensure balance in key clinical features thought to be related to outcome, subjects will be stratified into one of four categories based on the two main clinical features: nasal polyps (presence/absence) and history of previous sinus surgery (yes/no) prior to randomization.

Intervention The study intervention will be budesonide powder (0.5 mg/capsule) or an identical-appearing placebo product containing lactose. All subjects will be provided with the 8-ounce (240 ml) NeilMed Sinus Rinse Regular Bottle Kit and a one-month supply of USP Grade Sodium Chloride & Sodium Bicarbonate Mixture (pH balanced, Isotonic & Preservative & Iodine Free) commercially prepared packettes. Subjects may substitute the NeilMed Sinus Rinse Regular Bottle Kit for a nasal irrigation system, which in the opinion of the Principal Investigator, is similar to the NeilMed system and embodies the low-pressure, high-volume concept of nasal irrigation. Subjects will need to purchase distilled water or boil tap water for five minutes for use with the saline irrigation. Subjects will be required to dissolve the contents of two capsules into the 8-ounce (240 ml) NeilMed Sinus Rinse Regular Bottle along with the saline rinse. All subjects will be instructed to irrigate both right and left nasal cavity with one-half of the contents of the nasal rinse once daily. The subjects will receive written instructions and a video prior to initiation of the intervention to ensure proper delivery.

Each study bottle will contain 60 capsules of Budesonide or placebo and will be assigned with a number from 1-80. Only Dr. Kallogjeri (biostatistician) will have a list that links the treatment type (Budesonide or placebo) with the bottle number. The bottle number will correspond to the randomization schedule provided from Dr. Kallogjeri. The subject and the rest of the study team will remain blinded to the randomization assignment. The subject and the rest of the study team will only know what bottle number is being assigned, not which treatment is contained in each bottle. Dr. Kallogjeri is the biostatistician of the study and otherwise is not involved with the participants.

In the event of a Serious Adverse Event determined by the PI to necessitate the breaking of the blind, the intervention assignment will be revealed by Dr. Kallogjeri to the medical staff doctor caring for the patient. In the event Dr. Kallogjeri is unable to be reached in a time needed, to assure the safety of the subject, the blind can be broken by Sara Kukuljan, RN, or Drs. Piccirillo or Schneider and information will be shared with the medical staff assuming care for the patient.

The active drug and placebo will be prepared by Genesis Pharmacy, St. Louis Missouri and delivered to the Clinical Outcomes Office where the products will be stored in a locked cabinet. The cost of sufficient budesonide for the study duration (i.e., 60 budesonide capsules) will be $75 and the cost of sufficient quantity of lactose capsules will be $25.

Budesonide Budesonide is an anti-inflammatory glucocorticoid steroid that is used for a variety of common ailments. Among conditions related to the respiratory tract, budesonide is used as an inhalational drug for the treatment of asthma, COPD, allergic rhinitis, and nasal polyps. The mechanism of action of budesonide is similar to other corticosteroids and includes a wide range of inhibitory activities against multiple cell types (e.g., mast cells, eosinophils, neutrophils, macrophages and lymphocytes) and mediators (eg, histamine, eicosanoids, leukotrienes, and cytokines) involved in allergic- and non-allergic-mediated inflammation.(AstraZeneca 2000)

Subjects randomized to the budesonide intervention arm will be required to mix 1.0 mg (provided as two capsules containing 0.5 mg budesonide each) budesonide into the sinus rinse bottle and rinse each nasal cavity with one half of the bottle (~ 4 ounces or ~120 ml) daily. The inert ingredients are: loxasperse powder, which increases solubility and dispersibility of budesonide and is microbiologically safe; mannitol, which is widely used in pharmaceutical products as a capsule diluent; and Xylifos™ powder, which is a proprietary powder excipient used safely in pharmaceutical compounding for nasal nebulization or nasal irrigation.

Placebo The placebo product will contain lactose monohydrate and will be supplied in clear plastic capsules, which are identical to the budesonide capsules. The lactose capsule will only contain lactose as there are no other ingredients.

Concomitant Medications At the time of enrollment, most subjects will be expected to already be using topical nasal steroid medication (ie., fluticasone or Flonase®). Subjects currently using a topical nasal steroid spray will be asked to continue this medication. Topical nasal steroid sprays are indicated therapy for CRS and not considered experimental. Subjects not currently using a topical steroid spray will be asked to not initiate therapy during the duration of the study, unless there is a medical reason to use.

ELIGIBILITY:
Inclusion Criteria:

Twelve (12) weeks or longer of two or more of the following signs and symptom consistent with chronic rhinosinusitis (CRS)

• mucopurulent drainage (anterior, posterior, or both), nasal obstruction (congestion),facial pain-pressure-fullness, and decreased sense of smell

AND inflammation documented by one or more of the following findings:

* purulent (not clear) mucus or edema in the middle meatus or ethmoid region,
* polyps in nasal cavity or the middle meatus, and/or
* radiographic imaging showing inflammation of the paranasal sinuses

Exclusion Criteria:

* Unable to speak English
* History of comorbid ciliary dyskinesia, cystic fibrosis or any other mucociliary condition
* Dependence on prolonged corticosteroid therapy for comorbid conditions, such as asthma and chronic obstructive pulmonary disease.
* History of oral or systematic antibiotic use in the past 2 weeks
* History of nasal or sinus surgery within past 6 weeks
* History of cerebrospinal fluid leak
* History of allergy to budesonide or other topical steroids
* Pregnant or breast feeding
* Current infection or history of one of the following infections: Tuberculosis (TB) lung infection, or Herpes infection of the eye.
* Baseline SNOT-22 total scores below 9 were excluded due to the inability to achieve a minimally clinically improved difference

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-04-13 (Actual); Study Completion 2017-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay F Piccirillo, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Report of the Rhinosinusitis Task Force Committee Meeting. Alexandria, Virginia, August 17, 1996. Otolaryngol Head Neck Surg. 1997 Sep;117(3 Pt 2):S1-68. No abstract available. PMID 9380416
- [Background] Benninger MS, Ferguson BJ, Hadley JA, Hamilos DL, Jacobs M, Kennedy DW, Lanza DC, Marple BF, Osguthorpe JD, Stankiewicz JA, Anon J, Denneny J, Emanuel I, Levine H. Adult chronic rhinosinusitis: definitions, diagnosis, epidemiology, and pathophysiology. Otolaryngol Head Neck Surg. 2003 Sep;129(3 Suppl):S1-32. doi: 10.1016/s0194-5998(03)01397-4. No abstract available. PMID 12958561
- [Background] Snidvongs K, Pratt E, Chin D, Sacks R, Earls P, Harvey RJ. Corticosteroid nasal irrigations after endoscopic sinus surgery in the management of chronic rhinosinusitis. Int Forum Allergy Rhinol. 2012 Sep-Oct;2(5):415-21. doi: 10.1002/alr.21047. Epub 2012 May 7. PMID 22566474
- [Background] Sachanandani NS, Piccirillo JF, Kramper MA, Thawley SE, Vlahiotis A. The effect of nasally administered budesonide respules on adrenal cortex function in patients with chronic rhinosinusitis. Arch Otolaryngol Head Neck Surg. 2009 Mar;135(3):303-7. doi: 10.1001/archoto.2008.555. PMID 19289711
- [Background] Steinke JW, Payne SC, Tessier ME, Borish LO, Han JK, Borish LC. Pilot study of budesonide inhalant suspension irrigations for chronic eosinophilic sinusitis. J Allergy Clin Immunol. 2009 Dec;124(6):1352-4.e7. doi: 10.1016/j.jaci.2009.09.018. No abstract available. PMID 19910027
- [Background] Piccirillo JF, Merritt MG Jr, Richards ML. Psychometric and clinimetric validity of the 20-Item Sino-Nasal Outcome Test (SNOT-20). Otolaryngol Head Neck Surg. 2002 Jan;126(1):41-7. doi: 10.1067/mhn.2002.121022. PMID 11821764
- [Background] Browne JP, Hopkins C, Slack R, Cano SJ. The Sino-Nasal Outcome Test (SNOT): can we make it more clinically meaningful? Otolaryngol Head Neck Surg. 2007 May;136(5):736-41. doi: 10.1016/j.otohns.2007.01.024. PMID 17478207
- [Derived] Tait S, Kallogjeri D, Suko J, Kukuljan S, Schneider J, Piccirillo JF. Effect of Budesonide Added to Large-Volume, Low-pressure Saline Sinus Irrigation for Chronic Rhinosinusitis: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2018 Jul 1;144(7):605-612. doi: 10.1001/jamaoto.2018.0667. PMID 29879268
- Available data/document: Questionnaire: CGI scale — https://www.psywellness.com.sg/docs/CGI.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Men and women aged 18 and older with a diagnosis of chronic rhinosinusitis were recruited from the Washington University in St. Louis School of Medicine Otolaryngology clinic from January 1, 2016 to February 16, 2017.
Groups:
- Budesonide: The study intervention will be budesonide powder (0.5 mg/capsule). Subjects will be required to dissolve the contents of two capsules into the 8-ounce (240 ml) NeilMed Sinus Rinse Regular Bottle along with the saline rinse. All subjects will be instructed to irrigate both right and left nasal cavity with one-half of the contents of the nasal rinse once daily for 30 days..
  Each study bottle will contain 60 capsules of Budesonide and will be assigned with a number from 1-80.
  Budesonide: Participants will undergo 30-day treatment course that includes budesonide powder added to saline rinse.
- Saline Alone: Each study bottle will contain 60 capsules of placebo, which is lactose monohydrate and will be supplied in clear plastic capsules identical to the budesonide capsules. Subjects will be required to dissolve the contents of two capsules into the 8-ounce (240 ml) NeilMed Sinus Rinse Regular Bottle along with the saline rinse. All subjects will be instructed to irrigate both right and left nasal cavity with one-half of the contents of the nasal rinse once daily for 30 days.
  Saline alone: Participants will undergo 30-day treatment course that includes lactose (placebo) powder added to saline rinse.
Period: Overall Study
Arm/Group | Budesonide | Saline Alone
Started | 40 | 40
Completed | 29 | 32
Not Completed | 11 | 8
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Lost to Follow-up | 8 | 5

BASELINE CHARACTERISTICS:
Population: Study participants who completed intervention. Participants withdrawn from the study were excluded.
Groups:
- Total: Total of all reporting groups
Arm/Group | Budesonide | Saline Alone | Total
Number analyzed (Participants) | 37 | 37 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (14.1) | 48 (15.2) | 51 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 50
  Male | 12 | 12 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 33 | 34 | 67
  Race: African American | 3 | 2 | 5
  Race: Other | 1 | 1 | 2
Overall Comorbidity (ACE-27) [Count of Participants; unit: Participants] — ACE-27 measures the overall severity of comorbid ailments based on the degree of organ de-compensation (none, mild, moderate, or severe). The validated ACE-27 instrument lists various individual comorbid ailments and allows for the identification of degree of organ de-compensation for each ailment. Using a validated scoring method, the overall score of ACE-27 categorizes participants into 4 categories (0=None, 1=Mild, 2=Moderate, or 3=Severe) with category 0 presenting healthy participants with no comorbidities, and category 3 presenting the very sick participants.
  Participants
    None | 17 | 22 | 39
    Mild | 18 | 10 | 28
    Moderate | 2 | 3 | 5
    Severe | 0 | 2 | 2
Polyps [Count of Participants; unit: Participants]
  Yes | 12 | 6 | 18
  No | 23 | 31 | 54
  Unknown | 2 | 0 | 2
History of sinus surgery [Count of Participants; unit: Participants]
  Yes | 9 | 12 | 21
  No | 28 | 25 | 53
Baseline Endoscopic Score [Mean (Standard Deviation); unit: Scores on a scale] — The findings from the endoscopic examination will be collected using the grading system proposed by Lund and Kennedy.(Lund and Kennedy 1997). The LK Endoskopy grading system consits of five terms: Polyposis, discharge, edema, scarring, and crusting. Each of the five terms is graded on an ordinal scale ranging from 0 to 2, and are evaluated for each side of the nose. The Baseline Endoscopic Score is the sum of the scores (ranging from 0-20) with the higher scores indication worse disease.
  Scores on a scale | 5.8 (2.5) | 4.9 (1.9) | 5.3 (2.2)
Baseline SNOT-22 Total [Mean (Standard Deviation); unit: scores on a scale] — The SNOT-22 instrument includes a list of 22 symptoms and social/emotional consequences of rhinosinusitis. Each item is scored on a likert scale ranging from 0-5, with 0 being the best option (not a problem). The total score is calculated as the sum of individual items' responses and can range on a scale from 0-110, with higher scores reflecting worse physical problems, functional, limitations, and emotional characteristics due to chronic rhinosinusitis.
  scores on a scale | 43.4 (17.5) | 44.8 (19.7) | 44.1 (18.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in SNOT-22 (Sino-Nasal Outcome Test)
Description: The change in Sino-Nasal Outcome test (SNOT-22) scores between baseline and four weeks will serve as the primary outcome measure in this study and will be calculated as:
  Primary Outcome Measure, ∆SNOT-22 = SNOT-22 baseline - SNOT-22 4-week follow-up.
  The change in SNOT-22 score is measured on a scale from -110 to 110 with positive scores showing improvement with treatment and negative scores showing worse condition after treatment.
Time Frame: Baseline to 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Budesonide | Saline Alone
Number analyzed (Participants) | 29 | 32
score on a scale | 20.7 (17.9) | 13.6 (18.8)

2. Secondary Outcome: Clinical Global Impression of Change (CGI)
Description: The overall response to treatment will be measured with a modification of the Clinical Global Impression of change (CGI) scale. Upon completion of the study, subjects will be asked to answer the following question: "Overall, how would you rate your response to treatment?" Response options are: 1 = Very Much Improved, 2 = Much Improved, 3 = Minimally Improved, 4 = No Change, 5 = Minimally Worse, 6 = Much Worse, 7 = Very Much Worse. Higher scores mean worse response to treatment.
Time Frame: 4 weeks
Population: Reported counts of patients who self-reported "minimally improved," "much improved," or "very much improved"
Measure: Count of Participants; unit: Participants
Arm/Group | Budesonide | Saline Alone
Number analyzed (Participants) | 29 | 32
Participants | 24 | 20

3. Other Pre Specified Outcome: Change in Endoscopic Scores
Description: The change in Endoscopic Scores will be defined as the difference in the Lund-Kennedy Endoscopic score at baseline minus the Lund-Kennedy Endoscopic Score at 4 weeks and will be measured as the difference in scores on a scale that ranges from 0 to 20. Larger positive change reflects better response to treatment.
Time Frame: Baseline to 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Budesonide | Saline Alone
Number analyzed (Participants) | 29 | 32
score on a scale | 3.4 (2.3) | 2.7 (1.9)

ADVERSE EVENTS:
Time Frame: 8 weeks (4 weeks intervention and 4 weeks post-intervention)
Arm/Group | Budesonide | Saline Alone
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/32
Other Adverse Events (participants affected / at risk) | 0/29 | 0/32

LIMITATIONS AND CAVEATS:
The duration of the trial was only four weeks may have been an insufficient amount of time to see the complete effect of the budesonide therapy for chronic rhino-sinusitis. Compliance was assessed with patient self-reports.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-01): https://cdn.clinicaltrials.gov/large-docs/50/NCT02696850/Prot_SAP_000.pdf